CLINICAL TRIAL: NCT04204967
Title: Impact of Totally Transdermal Sedation in the Weaning From Remifentanil Infusion Among Critically Ill Patients Undergoing Mechanical Ventilation: a Pilot Randomized-controlled Study (The TOES Trial)
Brief Title: Totally Transdermal Sedation in the Weaning From Remifentanil Infusion
Acronym: TOES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2687; 2019-002509-22 (EudraCT Number)
Record Dates: First submitted 2019-12-07; First posted 2019-12-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Insufficiency; Ventilator Weaning; Analgesics, Opioid
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: 2-arm, single-center, prospective randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transdermal fentanyl (Experimental): transdermal fentanyl will be administered with a starting dose of 50 mcg/hr simultaneously with the preexistent remifentanil continue infusion. Remifentanil infusion rate will be increased or decreased based on PaCO2 value resulting from the Arterial Blood Gases sample (ABG) collected at each visit. After randomization, the transdermal fentanyl dose can be modified every 24 hours according to the study protocol to achieve the desired effect in terms of PaCO2 value resulting from the Arterial Blood Gases sample (ABG) collected
  Interventions: Drug: Fentanyl Transdermal System; Drug: Remifentanil
- IV Remifentanil alone (Active Comparator): remifentanil infusion is administered alone, the infusion rate will be increased or decreased according to the study protocol based on PaCO2 value resulting from the Arterial Blood Gases sample (ABG) collected at each visit
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Fentanyl Transdermal System — in the experimental arm transdermal fentanyl will be administered with a starting dose of 50 mcg/hr simultaneously with the preexistent remifentanil continue infusion. Remifentanil infusion rate will be increased or decreased based on PaCO2 value resulting from the Arterial Blood Gases sample (ABG) collected at each visit. After randomization, the transdermal fentanyl dose can be modified every 24 hours according to the study protocol to achieve the desired effect in terms of PaCO2 value resulting from the Arterial Blood Gases sample (ABG) collected
  Other Names: Alghedon
  Arms: transdermal fentanyl
Drug: Remifentanil — In the active comparator arm remifentanil infusion is administered alone, the infusion rate will be increased or decreased according to the study protocol based on PaCO2 value resulting from the Arterial Blood Gases sample (ABG) collected at each visit.
  In the experimental arm remifentanil is use together with transdermal fentanyl
  Other Names: Ultiva

SUMMARY:
The choice of the sedation protocol has a massive impact on the duration of mechanical ventilation and the timing of extubation. Many sedation protocols are described in the literature. The investigators aim to assess if a transdermal fentanyl-based sedation protocol can have an impact on the global Work of Breathing (WOB)

DETAILED DESCRIPTION:
The choice of the sedation protocol has a massive impact on the duration of mechanical ventilation and the timing of extubation. Many sedation protocols are described in the literature. No data are available about the possibility of using transdermal fentanyl as an alternative to intravenous opioids during the weaning phase from mechanical ventilation and the post-extubation period until the discharge from ICU to the ward. The investigators aim to assess if a transdermal fentanyl-based sedation protocol can have an impact on the global Work of Breathing (WOB). Secondary endpoints of the study are the duration of mechanical ventilation, the duration of continuous infusion of opioids, the length of stay in ICU and in hospital. Eligible patients will be randomized in 2 groups: Group 1 will receive remifentanil; Group 2 will receive transdermal fentanyl and remifentanil. An Edi Catheter for diaphragm electrical activity monitoring will be put in place for each patient.

Statistical Analysis: Distribution normality will be assessed with the Kolmogorov-Smirnov test. Continuous variables will be reported expressed as medians (interquartile ranges). Qualitative variables will be reported as frequencies. Analysis on the primary efficacy criterion and other quantitative variables will be assessed with the Wilcoxon-Mann-Whitney test. Categorical outcomes will be compared with the chi-square test, or Fisher's exact test, as appropriate. Cochran-Mantel-Haenszel statistics will be reported for all these results. Two-way analysis of variance (ANOVA) for repeated measures with Bonferroni correction will be used to determine the differences in secondary endpoints. Comparisons between groups regarding these variables at each study time point were performed with the Student's t-test or Mann-Whitney test, as appropriate. Mean difference and 95% confidence interval [Confidence Interval 95%] are reported for most significant results. Two-tail p values≤0.05 Will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yo;
* Negative pregnancy test prior to inclusion in the study;
* The informed consent form needs to be signed and dated by the patient or a relative/legal guardian before of any procedure related to the study; if the patient is initially unable to sign the informed consent form, but later regains the ability to sign it, a new informed consent form will be given to the patient and must be signed and dated;
* Mechanically ventilated in Pressure Support Ventilation, according to the decision to the attending physician;
* A patient with prolonged weaning from the mechanical ventilator will be considered eligible. Prolonged weaning is defined as weaning that is still not terminated 7 days after the first separation attempt from the ventilator (by success or death).
* Analgesia provided by continuous infusion of remifentanil lasting five days or more and an intolerance to a dose reduction of 0.025 mcg/kg/min defined as the presence of at least one of the following criteria: RASS ≥ 2, a respiratory rate ≥ 35 breaths/minute, a PaCO2 < 30 mmHg, a heart rate > 120 bpm, a systolic blood pressure value > 160 mmHg or an increase of Visual Analogue Scale for pain assessment of ≥ 2 points.

Exclusion Criteria:

* Hypersensitivity to the active substance or any of the excipients;
* Hepatic or renal impairment;
* Fever (body temperature ≥ 38 °C) or septic shock, hypothermia (body temperature < 35 °C) or presence of active surface cooling systems;
* Hypercapnic patients with a PaCO2 > 45 mmHg;
* Current enrollment or plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 30 days or 5 half-lives of the agent, prior to the baseline visit;
* Hypoxemic respiratory failure (P/F < 200 mmHg);
* Delirium state defined as RASS ≥ 3 and CAM-ICU positive;
* Hemodynamic instability requiring high doses of inotropes or vasopressors;
* Any condition that may contraindicate the use of remifentanil or transdermal fentanyl;
* Patients with a BMI ≥ 35;
* Patient admitted for postoperative monitoring after elective surgery;
* EAdi catheter contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the work of breathing (WOB) of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  To demonstrate that the area under the curve (AUC) of the work of breathing per minute (cmH20*sec/min) (assessed at 1, 6, 12, 24 hours for the first day after randomization, and every 24 hours for the following days) in the intervention group is not higher than the control group.
Comparison of the work of breathing per breath of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  cmH20*sec/min
Comparison of the inspiratory effort of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  cmH20
Comparison of the delta electrical activity of the diaphragm (EAdi) of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  microvolt (mcv)
Comparison of the plateau pressures of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  cmH20
Comparison of driving pressures of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  cmH20
Comparison of transpulmonary driving pressures of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  cmH20
Comparison of the pulmonary compliance of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  ml/cmH20
Comparison of P0.1 of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  cmH20
Comparison of P/F ratios of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  The P/F ratio equals the arterial PaO2 (Arterial Oxygen Partial Pressure) (mmHg) divided by the FIO2 (the fraction of inspired oxygen expressed as a decimal)

SECONDARY OUTCOMES:
Comparison of respiratory rates of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  breaths per minute
Comparison of tidal volumes of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  milliliters
Comparison of arterial blood pressure of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  mmHg
Comparison of heart rates of the patients randomized to receive transdermal fentanyl vs. remifentanil alone. | starts with the randomization and ends 72 hours after randomization
  bpm
Global duration of mechanical ventilation among the two groups. | starts with the randomization and ends with the discharge from the intensive care unit.
  Days
Global duration of intravenous remifentanil infusion among the two groups. | starts with the randomization and ends with the discharge from the intensive care unit.
  Hours
Length of stay in hospital among the two groups. | starts with the randomization and ends with the discharge from the Hospital.
  Days
Length of stay in ICU among the two groups. | starts with the randomization and ends with the discharge from the intensive care unit.
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. A Caricato, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong BH, Ko MG, Nam J, Yoo H, Chung CR, Suh GY, Jeon K. Differences in clinical outcomes according to weaning classifications in medical intensive care units. PLoS One. 2015 Apr 15;10(4):e0122810. doi: 10.1371/journal.pone.0122810. eCollection 2015. PMID 25876004
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Girard TD, Alhazzani W, Kress JP, Ouellette DR, Schmidt GA, Truwit JD, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Morris PE; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. An Official American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Rehabilitation Protocols, Ventilator Liberation Protocols, and Cuff Leak Tests. Am J Respir Crit Care Med. 2017 Jan 1;195(1):120-133. doi: 10.1164/rccm.201610-2075ST. PMID 27762595
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Perkins GD, Mistry D, Gates S, Gao F, Snelson C, Hart N, Camporota L, Varley J, Carle C, Paramasivam E, Hoddell B, McAuley DF, Walsh TS, Blackwood B, Rose L, Lamb SE, Petrou S, Young D, Lall R; Breathe Collaborators. Effect of Protocolized Weaning With Early Extubation to Noninvasive Ventilation vs Invasive Weaning on Time to Liberation From Mechanical Ventilation Among Patients With Respiratory Failure: The Breathe Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1881-1888. doi: 10.1001/jama.2018.13763. PMID 30347090
- [Background] Muellejans B, Lopez A, Cross MH, Bonome C, Morrison L, Kirkham AJ. Remifentanil versus fentanyl for analgesia based sedation to provide patient comfort in the intensive care unit: a randomized, double-blind controlled trial [ISRCTN43755713]. Crit Care. 2004 Feb;8(1):R1-R11. doi: 10.1186/cc2398. Epub 2003 Nov 20. PMID 14975049
- [Background] Akinci SB, Kanbak M, Guler A, Aypar U. Remifentanil versus fentanyl for short-term analgesia-based sedation in mechanically ventilated postoperative children. Paediatr Anaesth. 2005 Oct;15(10):870-8. doi: 10.1111/j.1460-9592.2005.01574.x. PMID 16176316
- [Background] Zhu Y, Wang Y, Du B, Xi X. Could remifentanil reduce duration of mechanical ventilation in comparison with other opioids for mechanically ventilated patients? A systematic review and meta-analysis. Crit Care. 2017 Aug 3;21(1):206. doi: 10.1186/s13054-017-1789-8. PMID 28774327
- [Background] Futier E, Chanques G, Cayot Constantin S, Vernis L, Barres A, Guerin R, Chartier C, Perbet S, Petit A, Jabaudon M, Bazin JE, Constantin JM. Influence of opioid choice on mechanical ventilation duration and ICU length of stay. Minerva Anestesiol. 2012 Jan;78(1):46-53. Epub 2011 Nov 5. PMID 21971434
- [Background] Natalini G, Di Maio A, Rosano A, Ferretti P, Bertelli M, Bernardini A. Remifentanil improves breathing pattern and reduces inspiratory workload in tachypneic patients. Respir Care. 2011 Jun;56(6):827-33. doi: 10.4187/respcare.01014. Epub 2011 Feb 11. PMID 21333087
- [Background] Newshan G. Heat-related toxicity with the fentanyl transdermal patch. J Pain Symptom Manage. 1998 Nov;16(5):277-8. doi: 10.1016/s0885-3924(98)00100-6. No abstract available. PMID 9846020
- [Background] Carter KA. Heat-associated increase in transdermal fentanyl absorption. Am J Health Syst Pharm. 2003 Jan 15;60(2):191-2. doi: 10.1093/ajhp/60.2.191. No abstract available. PMID 12561665
- [Background] Lotsch J, Walter C, Parnham MJ, Oertel BG, Geisslinger G. Pharmacokinetics of non-intravenous formulations of fentanyl. Clin Pharmacokinet. 2013 Jan;52(1):23-36. doi: 10.1007/s40262-012-0016-7. PMID 23100195
- [Background] Bulow HH, Linnemann M, Berg H, Lang-Jensen T, LaCour S, Jonsson T. Respiratory changes during treatment of postoperative pain with high dose transdermal fentanyl. Acta Anaesthesiol Scand. 1995 Aug;39(6):835-9. doi: 10.1111/j.1399-6576.1995.tb04180.x. PMID 7484044
- [Background] Beck J, Gottfried SB, Navalesi P, Skrobik Y, Comtois N, Rossini M, Sinderby C. Electrical activity of the diaphragm during pressure support ventilation in acute respiratory failure. Am J Respir Crit Care Med. 2001 Aug 1;164(3):419-24. doi: 10.1164/ajrccm.164.3.2009018. PMID 11500343
- [Background] Bellani G, Mauri T, Coppadoro A, Grasselli G, Patroniti N, Spadaro S, Sala V, Foti G, Pesenti A. Estimation of patient's inspiratory effort from the electrical activity of the diaphragm. Crit Care Med. 2013 Jun;41(6):1483-91. doi: 10.1097/CCM.0b013e31827caba0. PMID 23478659
- [Background] Liu L, Liu H, Yang Y, Huang Y, Liu S, Beck J, Slutsky AS, Sinderby C, Qiu H. Neuroventilatory efficiency and extubation readiness in critically ill patients. Crit Care. 2012 Jul 31;16(4):R143. doi: 10.1186/cc11451. PMID 22849707
- [Background] Jansen D, Jonkman AH, Roesthuis L, Gadgil S, van der Hoeven JG, Scheffer GJ, Girbes A, Doorduin J, Sinderby CS, Heunks LMA. Estimation of the diaphragm neuromuscular efficiency index in mechanically ventilated critically ill patients. Crit Care. 2018 Sep 27;22(1):238. doi: 10.1186/s13054-018-2172-0. PMID 30261920
- [Background] Adachi YU, Sano H, Doi M, Sato S. Central neurogenic hyperventilation treated with intravenous fentanyl followed by transdermal application. J Anesth. 2007;21(3):417-9. doi: 10.1007/s00540-007-0526-x. Epub 2007 Aug 1. PMID 17680198
- [Background] Delorme M, Bouchard PA, Simon M, Simard S, Lellouche F. Effects of High-Flow Nasal Cannula on the Work of Breathing in Patients Recovering From Acute Respiratory Failure. Crit Care Med. 2017 Dec;45(12):1981-1988. doi: 10.1097/CCM.0000000000002693. PMID 28857852
- [Background] Lellouche F, Maggiore SM, Deye N, Taille S, Pigeot J, Harf A, Brochard L. Effect of the humidification device on the work of breathing during noninvasive ventilation. Intensive Care Med. 2002 Nov;28(11):1582-9. doi: 10.1007/s00134-002-1518-9. Epub 2002 Oct 10. PMID 12415444

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT04204967/Prot_SAP_003.pdf